CLINICAL TRIAL: NCT00179790
Title: Reduced Intensity Stem Cell Transplant in Children and Young Adults Utilizing Photopheresis, Fludarabine, and Busulfan
Brief Title: Reduced Intensity Transplant Using Extracorporeal Photopheresis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Collaborators: Mallinckrodt (Industry)
Responsible Party: Principal Investigator, Jennifer Schneiderman, MD, Attending Physician, Hematology, Oncology,Cell Transplantation, Ann & Robert H Lurie Children's Hospital of Chicago
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ECP RIT
Record Dates: First submitted 2005-09-09; First posted 2005-09-16 (Estimated); Last update posted 2017-03-06 (Actual); Status verified 2017-03

CONDITIONS: Leukemia; Cancer
Keywords: cancer; hemoglobinopathy; immune deficiency; photopheresis; ECP; extracorporeal photopheresis
MeSH Terms: conditions — Leukemia; Neoplasms; Hemoglobinopathies; Immunologic Deficiency Syndromes | interventions — Photopheresis

INTERVENTIONS:
Procedure: Extracorporeal Photopheresis — Patient will undergo ECP treatment pre and post stem cell transplant infusion

SUMMARY:
Stem cell transplantation may be used to cure childhood cancers, and other diseases. Traditionally, stem cell transplants use high doses of chemotherapy and radiation. This regimen may cause significant problems after transplant such as infertility, infection, and graft versus host disease (GVHD).

Reduced intensity transplant (RIT) uses medications which weaken the immune system, allowing donor cells to take over. The goal of a RIT is to reduce the risk for complications after transplant. Usually medication is used to weaken the immune system, but there are other options such as extracorporeal photopheresis (ECP) that may be less toxic.

ECP is currently used for the treatment of GVHD and certain lymphomas. ECP uses a machine that filters white blood cells from the blood, treats them with ultraviolet (UV) light, and then gives all the cells back to the patient. The patient's immune system becomes weaker, allowing the donor cells to replace those of the patient. Studies involving the use of ECP for conditioning have shown fewer side effects than the use of medications.

The primary purpose of this clinical research trial is to evaluate the safety and feasibility of ECP as part of a preparative regimen for RIT in children and young adults.

DETAILED DESCRIPTION:
This study tests the feasibility of a reduced intensity preparative regimen for stem cell transplant including extracorporeal photopheresis (ECP), busulfan, and fludarabine in patients with leukemia, lymphoma, and certain non-malignant diseases. The current reduced intensity protocol includes busulfan, fludarabine, and anti-thymocyte immunoglobulin. ECP is currently used in diseases such as chronic GVHD and cutaneous T cell lymphoma. The mechanism of ECP has not been defined. It is hypothesized that exposure of white blood cells to ultraviolet light with 8-methoxypsoralen initiates an apoptotic cellular cascade. Apoptotic cells are recognized and removed by the reticuloendothelial system, initiating the secretion of anti-inflammatory cytokines and the reduction of proinflammatory cytokines. Antigen presenting cells then regulate immune responses through the induction of tolerance.

Here we incorporate the use of ECP, fludarabine, and busulfan in the preparative regimen, followed by ECP as prophylaxis for acute graft versus host disease. We hypothesize that photopheresis is safe and feasible, and patients will have similar rates of engraftment with less GVHD as those treated with current reduced intensity protocols. The use of ECP prior to transplant provides immunosuppression promoting host engraftment. Furthermore, the introduction of ECP following transplant may be able to induce tolerance thereby reducing rates of GVHD.

ELIGIBILITY:
Inclusion Criteria:

* Weight > 25 kg
* Patients with acute lymphoblastic leukemia (ALL) who are in CR (complete remission; < 5% blasts in bone marrow and no active central nervous system disease) who:

  * Are in second remission with an initial remission of < 36 months.
  * Patients with "high risk" disease in CR1, defined by karyotype abnormalities such as presence of (9;22) translocation, monosomy 7, or monosomy 5; and/or patients with slow initial response (initial remission not reached within four weeks from diagnosis).
  * Are in third (or subsequent) remission
  * Experience isolated extramedullary relapse while on therapy
  * Have experienced relapse following myeloablative stem cell transplant
  * Are WT1+ following induction therapy
* Patients with acute myelogenous leukemia (AML) who:

  * Are in first remission and remain WT1 positive.
  * Are in second remission
  * Are in initial partial remission (< 20% blasts in bone marrow)
  * Experience relapse following myeloablative stem cell transplant
* Patients with relapsed lymphoma whose residual disease appears to be chemo-responsive and non-bulky (< 5 cm largest diameter)
* Patients with chronic myelogenous leukemia (CML) in chronic phase who:

  * Don't achieve remission (molecular or cytogenetic) by 1 year of diagnosis with therapy (imatinib mesylate or interferon)
  * Have a rising quantitative bcr/abl on imatinib mesylate (molecular relapse)
  * Had developed accelerated phase regardless of therapy but are now back in second chronic phase
* Patients with recurrent solid tumors (neuroblastoma, Ewing's sarcoma, melanoma, rhabdomyosarcoma)
* Patients with myelodysplastic syndrome
* Patients with refractory anemia (RA) and refractory anemia with excess blasts (RAEB) are eligible, but refractory anemia with excess blasts in transformation (RAEB-T) patients are only eligible if treated to < 20% blasts with chemotherapy
* Patients with selected immunodeficiencies such as Wiskott-Aldrich syndrome or hyper-IgM syndrome
* Patients with metabolic diseases such as Niemann-Pick or adrenoleukodystrophy
* Patients with bone marrow failure syndromes, including aplastic anemia
* Adequate venous access

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2005-07; Primary Completion 2010-06 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
To determine the feasibility of using photopheresis as the backbone of a reduced intensity transplant regimen to reduce transplant related mortality and acute and chronic graft versus host disease (GVHD) | Throughout Treatment
To determine time to engraftment and the percentage of patients achieving full engraftment by day +100. Engraftment will be defined as > 95% total donor chimerism as determined by restriction fragment length polymorphism (RFLP). | By Day +100
To determine the rate of grades III and IV acute GVHD. | Throughout Treatment
To evaluate 100 day transplant related mortality | Through Day +100

SECONDARY OUTCOMES:
To establish patterns of biological effects of photopheresis on dendritic cell and CD4/CD8 populations, CD4/CD25 populations, IFN-gamma, TNF-alpha, IL-10, IL-12, and IL-4 | Pre Transplant through 1 year post stem cell transplant

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Schneiderman, MD, MS, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (1):
- Ann & Robert H Lurie Children's Hospital of Chicago, Chicago, Illinois, United States